CLINICAL TRIAL: NCT06826937
Title: Short Term Recall and Reprocess Therapy for PTSD
Brief Title: Short-Term Recall and Reprocess Therapy for Post Traumatic Stress Disorder (PTSD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ben-Gurion University of the Negev (Other)
Collaborators: Soroka University Medical Center (Other); Soroka Hospital,Beer Sheva,Israel (Unknown)
Responsible Party: Principal Investigator, Or Duek, Or Duek, PhD, Principal Investigator, Ben-Gurion University of the Negev
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SOR-24-0209
Record Dates: First submitted 2025-01-28; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: PTSD; Post Traumatic Stress Disorder
Keywords: Prolonged Exposure; Massed Therapy; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: People will be assigned to intervention or waiting list groups. The waiting list will be crossed over 3 months into the study (after the 90 follow-up point)
Who Masked: Outcomes Assessor
Masking Description: Data will be collected with group assignment masked. We will unmask the data for analysis in bulks of 20 patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reconsolidation based short term therapy (Experimental): This will include an intensive week-long intervention (see Duek et al., 2023). Following the first meeting with the therapist, in which life history will be taken, patients will meet on a daily basis for five consecutive days. During these days, the patient will undergo imaginal exposure followed by processing of the traumatic event. Later this day, the patient will undergo in-vivo exposure with a member of the research team.
  The patient will be followed up for up to five years.
  Interventions: Behavioral: Reconsolidation based short term therapy
- WaitList (No Intervention): Patients who will be randomized to this arm will start with no intervention (following the screening procedure). They will be monitored at the screening at 7, 30, and 90 days. After the last follow-up, crossover to the active group will be offered.

INTERVENTIONS:
Behavioral: Reconsolidation based short term therapy — This is a behavioral intervention that uses imaginal and in vivo exposure in daily meetings.
  Other Names: Short Term Recall and Reprocessing Therapy
  Arms: Reconsolidation based short term therapy

SUMMARY:
The goal of this clinical trial is to learn if a short-term behavioral intervention, based on imaginal and in-vivo exposure and psychodynamic reprocessing, works on alleviating Post-Traumatic Stress Disorder (PTSD) symptoms in adults. The trial will also learn about patterns of recovery and relapse by following the patients for up to five years. The main questions it aims to answer are:

Does the reconsolidation-based short-term intervention help alleviate PTSD symptoms? How is it affecting other mental health issues (such as depression, sleep problems, and general functioning)? What is the long-term effect of the intervention? Researchers will compare this behavioral intervention to a waiting list, for up to three months. People on the waiting list will then be able to cross over to the treatment arm as well.

Participants will:

Be screened by a clinical psychologist Take the week-long intensive behavioral intervention (psychotherapy) Followed at the end of treatment (day 7), at 30 and 90 days, and every 6 months, up to five years.

Wearable devices will be used during the week before treatment, during treatment, and up to 30 days following the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosis of PTSD with a score of 25 or higher (i.e. severe PTSD) on the Clinician- Administered PTSD Scale (CAPS-5) at screening.

  * Subjects on FDA-approved antidepressants, trazodone, atypical neuroleptic, prazosin, or clonidine may enter the study if they have been on a stable treatment, as determined by the study clinician, for at least 4 weeks prior to randomization. Following randomization, small changes to doses may be allowable at the PI's discretion.
  * Able to provide written informed consent.
  * Able to read and write English/Hebrew.

Exclusion Criteria:

* • Patients with a diagnostic history of bipolar disorder, borderline personality disorder, obsessive-compulsive disorder, schizophrenia or schizoaffective disorder or currently exhibiting psychotic features as determined by the clinical interview; dementia or suspicion thereof, are excluded. Other DSM Axis I disorders are permitted as long as they are not considered primary disorders.

  * Patients with a history of antidepressant-induced hypomania or mania as determined by open-ended psychiatric interview.
  * Current, ongoing serious suicidal risk as assessed by evaluating.
  * Moderate severity or greater Substance Use Disorder (excepting Alcohol Use Disorder) during the 3 months prior to randomization, as determined by the SCID.
  * History of traumatic brain injury (TBI) with loss of consciousness for more than 24 hours or posttraumatic amnesia for more than 7 days may be considered if the trauma occurred more than 1 year ago, and no more than minimal symptoms have persisted over the past year.
  * Any significant history of neurological illness or heart disease.
  * Any signs of major medical or neurological illness on examination or as a result of ECG screening or laboratory studies.
  * Any history indicating learning disability or mental retardation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in PTSD symptoms (PCL-5) | At screening, at the end of treatment (i.e., 7 days following the initiation of the treatment), at 30 days, at 90 days and up to 5 years follow-up (bi-annualy, i.e., every six months))
  Assessing changes in PTSD symptoms measured using the PTSD Checklist 5 (PCL-5). PCL uses a 5 point Likert scale ranging from "not at all" (0) to "extremely" (4). Score ranges between 0-80, with higher score means higher severity

SECONDARY OUTCOMES:
Improved sleep | 6 weeks total. One week before the beginning of the treatment, during treatment and up to 30 days follow-up.
  Sleep will be measured using both a self-report questionnaire and a Garmin Vivosmart 5 watch. This will include total sleep per day, average weekly (hours), and REM/total sleep time ratio. All will be measured using the wearable watch.
Depressive symptoms | At screening, at the end of treatment (i.e., 7 days following the initiation of the treatment), at 30 days, at 90 days and up to 5 years follow-up (bi-annualy, i.e., every six months))
  Depressive symptoms will be measured using the Beck Depression Inventory (BDI-II). Participants respond to each item using a 4-point Likert scale, ranging from 0 (not present) to 3 (severe), which allows for the quantification of symptom severity. Higher score corresponds to higher severity of depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Ben Gurion University of the Negev, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: Undecided
IPD is planned to be shared following a specific request and after identification.